CLINICAL TRIAL: NCT05963815
Title: Spine Patient Reported Outcome Measures: a Cohort Observational Study
Brief Title: The Spine PROMCO Study
Acronym: Spine PROMCO
Status: Recruiting | Type: Observational
Sponsor: Park Medical centrum (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0000090
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Disc Herniation; Spondylolisthesis; Spinal Stenosis
Keywords: Patient related outcome measures; Prognosis; Degenerative Spine disease
MeSH Terms: conditions — Intervertebral Disc Displacement; Spondylolisthesis; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Degenerative spine disorder: Patients who are eligible for surgical treatment of the spine, including a lumbar herniated disk or lumbar spinal canal stenosis, discopathy and spondylolisthesis.
  Interventions: Other: Spine surgery

INTERVENTIONS:
Other: Spine surgery — Patients operated with laminectomy, microscopic discectomy, percutaneous transforaminal endoscopic discectomy, and spondylodesis.

SUMMARY:
Our primary objective is to design a cohort to determine the treatment outcome of different surgical interventions of the degenerative lumbar spine highlighting the expediency and value of the current surgical treatment program.

DETAILED DESCRIPTION:
This observational prospective unicenter cohort study includes patients who are eligible for elective lumbar spine surgery due to a degenerative spine disease (e.g. herniated disk, spinal canal stenosis, discopathy and spondylolisthesis). An enrolment rate of at least 80% is pursued within minimal 1.5 years of inclusion. A digital survey is used including self-reporting questionnaires that pertain to outcomes as pain, functionality and disability (COMI Back), health status (EQ-5D-5L), re-operations and complications, and satisfaction. The survey is sent at given time-intervals (e.g. baseline 2 weeks prior to surgery, 6 weeks post surgery and 6, 12, 36 months post surgery). Besides descriptive statistics and multivariate analysis, an economic evaluation will be performed from a societal perspective.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are eligible for elective surgery of the lumbar spine.
* All patients with degenerative disorder of the lumbar spine including: herniated disk, stenosis, discopathy and spondylolisthesis.
* Patients must be able to fill in the questionnaire online
* Patients with imaging (Magnetic resonance imaging (MRI)) confirmed lumbar disc herniation, stenosis, discopathy, or listhesis.
* Elective cases
* Patients operated with laminectomy, microscopic discectomy, percutaneous transforaminal endoscopic discectomy, and spondylodesis.

Exclusion Criteria:

* Patients who cannot speak nor read the Dutch language
* Patients who are not able to complete the digital questionnaires, according to the including doctor
* Patients with fractures, primary infections of the spine, or with spinal malignant- cies.
* Patients in a traumatic setting.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible for surgical treatment of the spine, including a lumbar herniated disk or lumbar spinal canal stenosis, discopathy and spondylolisthesis.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2030-01-13 (Estimated); Study Completion 2030-01-13 (Estimated)

PRIMARY OUTCOMES:
Pain and functionality - COMI BACK | Baseline preoperative (about 2 weeks pre surgery). After completing the baseline measurements, the patients are asked to repeat the survey post surgery on set dates; 6 weeks-6months-12months-24 months-and 36 months post surgery
  The Core Outcome Measures Index (COMI) Back index score (range 0-10) is calculated by averaging transformed core-item scores from each domain of the five domains: pain symptoms (including NRS-scale), functionality of back, symptom-specific well-being, general well-being, and disability. Although the Oswestry disability index (ODI) is the most commonly used and cited tool, the COMI Back was chosen instead to assess pain intensity, functionality and disability within the study group. The COMI back is relatively short (7 questions), includes the NRS-scale (painscore from 0 (no pain) - 10 (worst possible pain), and has been cross-culturally adapted and validated in several languages, including in Dutch. It is the preferred tool of the Eurospine Registry.
Health status - EQ5DL | Baseline preoperative (about 2 weeks pre surgery). After completing the baseline measurements, the patients are asked to repeat the survey post surgery on set dates; 6 weeks-6months-12months-24 months-and 36 months post surgery
  The eq-5D-5L (Euroquality 5 domains 5 level) health questionnaire provides a simple descriptive profile and a single index value for health status. The EQ-VAS is part of the EQ-5D-5L and it is a visual scale in which the patient can indicate the perception of their health status at the time of assessment, with 100 being perfect health status and 0 the worst health status. With the EQ-5D-5L we can assess the quality-adjusted life years (QALY).

SECONDARY OUTCOMES:
Number of Re-operations | post surgery on set dates; 6 weeks-6months-12months-24 months-and 36 months post surgery
  Re-operation due to a complication or recidive is self-reported and registered in the Electronic medical record.
Complication | post surgery on set dates; 6 weeks-6months-12months-24 months-and 36 months post surgery
  Complications are systematically assessed by self-reported questionnaires (e.g. Cerebro spinal fluid leakage, sensomotoric deficits, incontinence, infections, etc).
Satisfaction | 6 weeks, 6-12-36 months post surgery
  Patient's satisfaction will be assessed using a 5-point Likert Scale to touch on the subject of: (1) hospital satisfaction, (2) treatment satisfaction, (3) recovery satisfaction and (4) response burden of the study. With 1 being very dissatisfied and 5 very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Park Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Parenteau CS, Lau EC, Campbell IC, Courtney A. Prevalence of spine degeneration diagnosis by type, age, gender, and obesity using Medicare data. Sci Rep. 2021 Mar 8;11(1):5389. doi: 10.1038/s41598-021-84724-6. PMID 33686128
- [Background] Konstantinou K, Dunn KM. Sciatica: review of epidemiological studies and prevalence estimates. Spine (Phila Pa 1976). 2008 Oct 15;33(22):2464-72. doi: 10.1097/BRS.0b013e318183a4a2. PMID 18923325
- [Background] Grotle M, Smastuen MC, Fjeld O, Grovle L, Helgeland J, Storheim K, Solberg TK, Zwart JA. Lumbar spine surgery across 15 years: trends, complications and reoperations in a longitudinal observational study from Norway. BMJ Open. 2019 Aug 1;9(8):e028743. doi: 10.1136/bmjopen-2018-028743. PMID 31375617
- [Background] Guzman JZ, Cutler HS, Connolly J, Skovrlj B, Mroz TE, Riew KD, Cho SK. Patient-Reported Outcome Instruments in Spine Surgery. Spine (Phila Pa 1976). 2016 Mar;41(5):429-37. doi: 10.1097/BRS.0000000000001211. PMID 26571179
- [Background] Asher AL, Knightly J, Mummaneni PV, Alvi MA, McGirt MJ, Yolcu YU, Chan AK, Glassman SD, Foley KT, Slotkin JR, Potts EA, Shaffrey ME, Shaffrey CI, Haid RW, Fu KM, Wang MY, Park P, Bisson EF, Harbaugh RE, Bydon M. Quality Outcomes Database Spine Care Project 2012-2020: milestones achieved in a collaborative North American outcomes registry to advance value-based spine care and evolution to the American Spine Registry. Neurosurg Focus. 2020 May 1;48(5):E2. doi: 10.3171/2020.2.FOCUS207. PMID 32357320
- [Background] van Hooff ML, Jacobs WC, Willems PC, Wouters MW, de Kleuver M, Peul WC, Ostelo RW, Fritzell P. Evidence and practice in spine registries. Acta Orthop. 2015;86(5):534-44. doi: 10.3109/17453674.2015.1043174. PMID 25909475
- [Background] Gadjradj PS, Chin-See-Chong TC, Donk D, Depauw P, Tulder MWV, Harhangi BS. Cross-Cultural Adaptation and Psychometric Validation of the Dutch Version of the Core Outcome Measures Index for the Neck in Patients Undergoing Surgery for Degenerative Disease of the Cervical Spine. Neurospine. 2021 Dec;18(4):798-805. doi: 10.14245/ns.2142682.341. Epub 2021 Dec 31. PMID 35000334
- [Background] Mannion AF, Vila-Casademunt A, Domingo-Sabat M, Wunderlin S, Pellise F, Bago J, Acaroglu E, Alanay A, Perez-Grueso FS, Obeid I, Kleinstuck FS; European Spine Study Group (ESSG). The Core Outcome Measures Index (COMI) is a responsive instrument for assessing the outcome of treatment for adult spinal deformity. Eur Spine J. 2016 Aug;25(8):2638-48. doi: 10.1007/s00586-015-4292-4. Epub 2015 Oct 30. PMID 26519374
- [Background] Devlin NJ, Brooks R. EQ-5D and the EuroQol Group: Past, Present and Future. Appl Health Econ Health Policy. 2017 Apr;15(2):127-137. doi: 10.1007/s40258-017-0310-5. PMID 28194657